CLINICAL TRIAL: NCT00169585
Title: A National, Multicentric, Randomised, Controlled Trial. Applications of a Critical Pathway Using Levofloxacin for the Management of Patients With Abnormal PSA.
Brief Title: Levofloxacin For The Management Of Patients With Abnormal Prostate Specific Antigen (PSA)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: LEV102341
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Prostatic Hyperplasia; Prostatitis
Keywords: diagnostic-therapeutic pathway; PSA; DRE; Levofloxacin
MeSH Terms: conditions — Prostatic Hyperplasia; Prostatitis | interventions — Levofloxacin

INTERVENTIONS:
Drug: Levofloxacin oral tablets

SUMMARY:
Multicentric, national, prospective, parallel group, controlled. The Subjects in every center will be randomized and assigned to the pharmacologic arm or the one with the biochemical monitoring

ELIGIBILITY:
Inclusion Criteria:

Only subjects who meet all of the following criteria will be eligible to participate in this study:

* Male patients
* Age ≥ 45 years
* Suspected presence of prostate inflammatory foci, defined according to the following criteria:
* PSA ≥ 2.6 ng/mL and age ≥ 50 and < 60 years (or ≥ 45 years if the patient has known family predisposition to carcinoma of the prostate) or,
* PSA ≥ 4.1 ng/mL and age ≥ 60 and < 75 years, and
* normal digito-rectal examination (DRE) (see section 5.2), and normal urine test with dipstick and/or microscopy carried out within 5 days of the baseline visit
* Patients willing and able to provide their written informed consent and to comply with study procedures.

  * Patients with LUTS/BPH on watchful waiting or already under treatment with alpha-blockers or 5-ARI (5-alpha reductase inhibitors) for at least 6 months will also be considered eligible to participate in the study.

Exclusion Criteria:

Patients who meet any of the following criteria will not be eligible to participate in this study:

* Diagnosis of NIH class I-III prostatitis or clinical evidence of active acute urinary infection and/or known or suspected active bacterial infection at other sites;
* Diagnosis of prostate carcinoma (or PIN or ASAPS) or prior radical prostatectomy or radiotherapy or other treatments for prostate cancer;
* PSA > 20 ng/mL;
* PSA values (including high values) stable over time;
* Start of a pharmacological therapy with 5-ARI in subjects with LUTS/BPH;
* Permanent catheter;
* Prior treatment (within 4 weeks) with levofloxacin for genital-urinary infections;
* Known or suspected allergy to levofloxacin, including the excipients contained in the pharmacological preparation and/or confirmed tendency to photosensitivity reactions after fluoroquinolone therapy;
* Concomitant treatment with drugs not allowed in the study
* Reluctance to undergo prostate biopsy and/or risk of non-compliance;
* History or current evidence of alcohol or drug abuse in the last 12 months;
* History of any conditions that, in the opinion of the investigator, may confound the study results or create additional risks for the patient.
* Participation in any study of investigational or marketed drugs within 30 days before the baseline visit or during the study.

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2005-03; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
To evaluate if the application of 3 weeks treatment of levofloxacin, compared with the execution of a prostatic biopsy, after biochemical monitoring of total PSA, could decrease significantly the level of serum concentration of total PSA in 6-7 weeks. | 6/7 week after treatment

SECONDARY OUTCOMES:
Normalization of serum concentration of total PSA; Changes in the time of levels of total PSA concentrations; Impact on patients''Qol(Quality of Life); Costs associated to both choices. | 24 weeks (follow-up visit)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MD, Study Director — GlaxoSmithKline
Locations (16):
- Italy (16):
  - GSK Investigational Site, Bari, Apulia
  - GSK Investigational Site, Foggia, Apulia
  - GSK Investigational Site, Matera, Basilicate
  - GSK Investigational Site, Avellino, Campania
  - GSK Investigational Site, Napoli, Campania
  - GSK Investigational Site, Bologna, Emilia-Romagna
  - GSK Investigational Site, Rome, Lazio
  - GSK Investigational Site, Lecco, Lombardy
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Lanzo Torinese (TO), Piedmont
  - GSK Investigational Site, Orbassano (TO), Piedmont
  - GSK Investigational Site, Turin, Piedmont
  - GSK Investigational Site, Sassari, Sardinia
  - GSK Investigational Site, Catania, Sicily
  - GSK Investigational Site, Messina, Sicily
  - GSK Investigational Site, Bagno A Ripoli (FI), Tuscany